CLINICAL TRIAL: NCT06169527
Title: French Prospective Observational Study of Patients Receiving Dupilumab for Atopic Dermatitis.
Brief Title: A Long-term Data Collection Study of Participants in France Aged 6 Years Old or More With Atopic Dermatitis Receiving Dupilumab
Acronym: DUPILAB
Status: Active, not recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS17668; U1111-1279-3469 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with AD treated with dupilumab: Patients ≥6 years of age in whom dupilumab therapy was initiated to treat their AD according to French-specific prescribing information.
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — Dupilumab cohort
  Other Names: SAR231893; Dupixent®

SUMMARY:
This is a long-term study to collect data over 3 years in order to find out what is likely to happen in the future regarding participants 6 years of age and older who receive dupilumab for Atopic Dermatitis (AD) commonly known as Eczema, and to characterize real-world effectiveness, safety and use patterns of dupilumab in real world setting in France. Patients will be invited to participate if initiating treatment with dupilumab for AD according to French-specific prescribing information. The decision of initiation of the treatment is independent to the study's participation. The study will be conducted in approximately 50 centers in France to evaluate a representative sample of patients treated in France. At each participating site, all AD participants who receive an initial prescription for dupilumab will be invited to participate in this study, until the enrollment goal is achieved.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 6 years or older.
* Initiating treatment with dupilumab for AD according to French-specific prescribing information (≥ 12 years old: moderate to severe AD versus 6-11 years old: severe AD). The decision of initiation of the treatment is independent to the study's participation.
* Able to understand and complete study-related questionnaires.
* Signed informed consent form. For participants <18 years old, Informed consent form signed by the parent/legal guardian and participant's assent obtained.

Exclusion Criteria:

* Patients who have a contraindication to the drug according to the French-specific prescribing information label.
* Any condition that, in the opinion of the Investigator, may interfere with patient's ability to participate in the study, such as short life expectancy, substance abuse, severe cognitive impairment, or other comorbidities that can predictably prevent the patient from adequately completing, as per routine care, the schedule of visits and assessments.
* Patients currently participating in any interventional clinical trial.
* Patients previously treated with dupilumab.
* Patients under tutorship or curatorship; patients under safeguard of justice or deprived of his/her liberty by an administrative or court decision.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population of interest for this study will be patients in France aged 6 years old or more with a diagnosis of AD either severe or moderate to severe (depending on age group) who initiate dupilumab in real world setting. The study will be conducted in real conditions of practice, dupilumab will be prescribed at the sole initiative of the participating physician irrespective of patient enrolment decision.
Sampling Method: Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2028-05-10 (Estimated); Study Completion 2028-05-10 (Estimated)

PRIMARY OUTCOMES:
Demographic characteristics of participants who receive dupilumab for AD | At baseline
  Including age, gender, educational level, socio-professional category
Weight characteristics of participants who receive dupilumab for AD | At baseline
Height characteristics of participants who receive dupilumab for AD | At baseline
Medical history characteristics of participants who receive dupilumab for AD | At baseline
  including previous treatments for AD, relevant medical history, family history of atopy
Comorbidities and treatments change from baseline | At baseline, month 3, month 6, month 12, month 18, month 24, month 30, month 36
Atopic comorbidities and treatments change from baseline | At baseline, month 3, month 6, month 12, month 18, month 24, month 30, month 36
Change from baseline in lifestyle habits of participants who receive dupilumab for AD | At baseline, month 3, month 6, month 12, month 18, month 24, month 30, month 36 if applicable
  Including alcohol, tobacco, CBD and cannabis consumption
Change from baseline in dupilumab dose | At baseline, month 3, month 6, month 12, month 18, month 24, month 30, month 36
Change from baseline in dupilumab administration | At baseline, month 3, month 6, month 12, month 18, month 24, month 30, month 36
Change from baseline in dupilumab compliance with treatment | At baseline, month 3, month 6, month 12, month 18, month 24, month 30, month 36
Change from baseline in dupilumab temporary or permanent discontinuation | At baseline, month 3, month 6, month 12, month 18, month 24, month 30, month 36
Change from baseline in dupilumab treatment switch to another therapy | At baseline, month 3, month 6, month 12, month 18, month 24, month 30, month 36
Change from baseline in dupilumab treatment for concomitant AD treatments | At baseline, month 3, month 6, month 12, month 18, month 24, month 30, month 36
Change in patient's treatment satisfaction score using the Patient Global Assessment of Treatment Effect (PGATE) | At month 6, month 12, month 18, month 24, month 30, month 36
  PGATE for patients ≥ 12 years of age: an internally developed and validated instrument allowing patients to rate their opinion and perceived treatment effect. Ratings are on a 5-point Likert scale from 1 being "Poor" and 5 being "Excellent".
Change in eczema severity using the Eczema Area and Severity Index (EASI) | At baseline, month 6, month 12, month 18, month 24, month 30, month 36
  EASI is a validated measure used to assess severity and extent of AD at each body region by multiplying the lesions characteristics score x the body area score x multiplier. Four AD disease characteristics -erythema, thickness (induration, population, and oedema), scratching (excoriation), and lichenification - will each be assessed for severity by the observing physician, as follows: 0 = none, absent; 1=mild (just perceptible); 2=Moderate (obvious); 3=Severe. The area score ranges from 0 to 6 is determined as follows: 0= 0% (no active eczema in region); 1= 1-9%; 2= 10-29%; 3= 30-49%; 4= 50-69%; 5= 70-89%; 6= 90-100% (entire region affected by eczema). The multiplier is determined according to the region affected and the age of the patient: 0.1 or 0.2 for patients < 8 years old (head/neck), 0.2 (upper limbs), 0.3 (trunk), 0.4 or 0.3 for patients < 8 years old (lower limbs). A higher score means higher AD severity. Scores range from 0 (no disease) to 72 (maximal disease severity).
Change in AD disease control using the Atopic Dermatitis Control Tool (ADCT) | At baseline, month 6, month 12, month 18, month 24, month 30, month 36
  ADCT for patients aged ≥ 12 years of age: a validated, brief and easily scored tool consisting of six concise questions allowing to rate the different dimensions of patient-perceived AD control, to foster communication between patients and their physicians and help appropriate decision-making. The instrument includes 6 items, with a 7-day recall period: overall severity of symptoms, frequency of intense episodes of itching, severity of bother, frequency of sleep impact, severity of daily activities impact and severity of mood or emotions impact. Each item is rated on a 5-point Likert scale, ranging from 0 (none/ not at all/ no nights) to 4 (very severe/ everyday/ extremely/ every night); the total score ranges from 0 to 24, which is the summation of the responses to all the items. A total score of ≥7 points was derived as the threshold to identify patients "not in control", based on optimal sensitivity/ specificity values. The higher the score, the less AD is controlled.
Change in itch assessment | At baseline, month 6, month 12, month 18, month 24, month 30, month 36
  Itch assessment (Worst-Itch Numeric Rating Scale, WI-NRS) will be rated from 0 to 10 on average during the past 7 days (adult, pediatric and adolescent patients), completed by the observing physician after questioning of patient; 0 = no itch and 10 = the worst imaginable itch.
Change in sleep disturbance NRS | At baseline, month 6, month 12, month 18, month 24, month 30, month 36
  NRS sleep disturbance will be rated from 0 to 10 on average during the past 7 days (adult, pediatric and adolescent patients), completed by the observing physician after questioning of patient; 0 = "sleep not disturbed at all" (best possible sleep) and 10 = "sleep extremely disturbed (worst possible sleep)".
Change in global patient's disease evaluation using the Patient Global Assessment of Disease Severity (PGADS) | At baseline, month 6, month 12, month 18, month 24, month 30, month 36
  PGADS for patients ≥ 12 years of age: an internally developed and validated instrument allowing to the patients to rate their AD-related overall well-being. Patients will be asked: "Considering all the ways in which your eczema affects you, how well are you doing?" Response choices will be from 1 being "Poor" to 5 being "Excellent".
Change in global patient's disease evaluation using the Caregiver Global Assessment of Disease (CGAD) | At baseline, month 6, month 12, month 18, month 24, month 30, month 36
  CGAD for patients 6 to 11 years of age: an internally developed and validated instrument allowing to the caregivers to rate their child's AD-related overall well-being. Caregivers will be asked: "Considering all the way in which the eczema affects your child, how well is your child doing?". Response choices will be 1 being "Poor" to 5 being "Excellent".
Change in Dermatology Life Quality Index (DLQI) | At baseline, month 6, month 12, month 18, month 24, month 30, month 36
  DLQI for patients ≥ 16 years (or cDLQI for patients < 16 at baseline) are 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on quality of life in adults and pediatrics, respectively. The format is a simple response (0 to 3 where 0 is "not at all" and 3 is "very much") to 10 items, which assess quality of life over the past week, with an overall scoring system of 0 to 30; a high score is indicative of a poor quality of life. Patients 6-11 years old will be assisted for questionnaire completion. A cDLQI's cartoon version could be also used for patients from 6 to 11 years old. If a patient turns 16 years old during the study, they will switch to DLQI.
Change in Dermatitis Family Impact Questionnaire (DFI) | At baseline, month 6, month 12, month 18, month 24, month 30, month 36
  DFI is a 10-item, validated questionnaire assessing the impact of AD on the QoL of the parents/legal representatives and family members of affected children. The format is a simple response (0 to 3 where 0 is "not at all" and 3 is "very much") to 10 items, which assess Quality of Life (QoL) over the past week, with an overall scoring system of 0 to 30; a high score is indicative of a poor QoL. It is designed to be completed by adults (aged 16 years or over) who have a child (up to and including the age of 15 years 11 months) in the family with atopic dermatitis.
Change in European Quality of Life-5 Dimensions-3 level score (EQ-5D-3L) | At baseline, month 6, month 12, month 18, month 24, month 30, month 36
  The EQ-5D-3L is completed by patients≥18 years old and by parent/legal representative of patients<18 years old. It consists of 2 parts:
  * The EQ-5D descriptive system has five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each has 3 levels: no problems, some problems, and extreme problems. The patient selects the most appropriate statement in each of the five dimensions, resulting in a 1-digit number for each dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  * The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement. The scale is numbered 0 to 100. A higher value represents better health and a lower value represents worse health.
Change in Work Productivity and Activity Impairment Questionnaire, Atopic Dermatitis (WPAI-AD) | At month 6, month 12, month 18, month 24, month 30, month 36
  WPAI-AD for adults and WPAI-CIQ-AD for adolescents is a questionnaire designed to assess the impact of AD on the patient's productivity. The WPAI-AD is the version of the original generic WPAI that is specific to AD. It is a 6-item, validated questionnaire to measure impairments in work and activities over a 7-day recall period. The WPAI-AD outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity. If a patient turns 18 years old during the study, this one will switch to WPAI-AD.
Number of Adverse Events (AE) | At baseline, month 3, month 6, month 12, month 18, month 24, month 30, month 36
  AEs for dupilumab and/or concomitant treatments will be collected throughout the study.
Change from baseline in Drug Survival | At baseline, month 3, month 6, month 12, month 18, month 24, month 30, month 36
  Drug survival is defined as the time from the start of treatment to the end or discontinuation of treatment with no changes. If a patient has multiple drug survival events for the same treatment, the longest drug survival will be used in the data summarization. The drug survival will be illustrated using a Kaplan-Meier plot.

CONTACTS AND LOCATIONS:
Locations (42):
- France (42):
  - Investigational Site Number: 2500041, Amiens
  - Investigational Site Number: 2500037, Angers
  - Investigational Site Number: 2500021, Argenteuil
  - Investigational Site Number: 2500044, Armentières
  - Investigational Site Number: 2500018, Arras
  - Investigational Site Number: 2500011, Ars-Laquenexy
  - Investigational Site Number: 2500023, Avignon
  - Investigational Site Number: 2500001, Besançon
  - Investigational Site Number: 2500003, Bron
  - Investigational Site Number: 2500043, Caen
  - Investigational Site Number: 2500050, Chambéry
  - Investigational Site Number: 2500006, Clermont-Ferrand
  - Investigational Site Number: 2500005, Dijon
  - Investigational Site Number: 2500004, Epagny Metz Tessy
  - Investigational Site Number: 2500039, Fort-de-France
  - Investigational Site Number: 2500045, La Tronche
  - Investigational Site Number: 2500019, Le Havre
  - Investigational Site Number: 2500040, Le Mans
  - Investigational Site Number: 2500038, Les Sables-d'Olonne
  - Investigational Site Number: 2500048, Levallois-Perret
  - Investigational Site Number: 2500032, Lille
  - Investigational Site Number: 2500002, Limoges
  - Investigational Site Number: 2500036, Lorient
  - Investigational Site Number: 2500029, Marseille
  - Investigational Site Number: 2500028, Montpellier
  - Investigational Site Number: 2500024, Nantes
  - Investigational Site Number: 2500025, Nice
  - Investigational Site Number: 2500020, Nice
  - Investigational Site Number: 2500016, Pau
  - Investigational Site Number: 2500009, Périgueux
  - Investigational Site Number: 2500042, Poitiers
  - Investigational Site Number: 2500022, Pontoise
  - Investigational Site Number: 2500014, Romans-sur-Isère
  - Investigational Site Number: 2500008, Rouen
  - Investigational Site Number: 2500015, Saint-Germain-en-Laye
  - Investigational Site Number: 2500027, Saint-Mandé
  - Investigational Site Number: 2500026, Saint-Nazaire
  - Investigational Site Number: 2500035, Saint-Pierre
  - Investigational Site Number: 2500013, Saint-Pierre
  - Investigational Site Number: 2500012, Toulouse
  - Investigational Site Number: 2500010, Valence
  - Investigational Site Number: 2500031, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org